CLINICAL TRIAL: NCT01619371
Title: Engorgement Study With the Simplisse Double Electric Breast Pump
Brief Title: Engorgement Study With a Double Electric Breast Pump
Status: Completed | Type: Observational
Sponsor: Foundation for Maternal Infant and Lactation Knowledge (Other)
Responsible Party: Sponsor
Other Study IDs: 2614
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Engorgement
Keywords: breast pump; engorgement; lactation
MeSH Terms: conditions — Hyperemia; Breast Milk Expression; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lactating women: Lactating women willing to use a breast pump.
  Interventions: Device: Simplisse Double Electric Breast Pump

INTERVENTIONS:
Device: Simplisse Double Electric Breast Pump — Use of breast pump for 10 minutes.
  Other Names: Simplisse Double Electric Breast Pump, 1005S

SUMMARY:
The purpose of this study is to analyze the effectiveness of an FDA approved Class II medical device, the Simplisse Double Electric Breast Pump, in relieving the symptoms of engorgement.

ELIGIBILITY:
Inclusion Criteria:

* first week postpartum seeking lactation management assistance for engorgement, identified as clinically engorged by health care practitioner.

Exclusion Criteria:

* greater than one week postpartum
* less than 18 years of age
* non-English speakers
* not willing to use double electric breast pump

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First 20 women arriving at the Newborn Care Center clinic in Reno, Nevada during their first week postpartum seeking lactation management assistance for engorgement.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Engorgement Relief | 10 minutes per subject
  Relief of engorgement as measured by the engorgement scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jimi Francis, MS,PhD,IBCLC, Principal Investigator — Foundation for Maternal Infant and Lactation Knowledge
Locations (1):
- Newborn Care Center Clinic, Reno, Nevada, United States

REFERENCES:
- See also: home page of sponsoring foundation — http://www.foundation4milk.org